CLINICAL TRIAL: NCT04189744
Title: Effects of Metronidazole Plus Intermittent Preventive Treatment of Malaria in Pregnancy on Birth Outcomes: a Randomised Controlled Trial in Zambia
Brief Title: The ASPIRE Trial - Aiming for Safe Pregnancies by Reducing Malaria and Infections of the Reproductive Tract
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ITDCZO83
Record Dates: First submitted 2019-10-28; First posted 2019-12-06 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-03

CONDITIONS: Pregnancy Malaria; Bacterial Vaginoses; Trichomonas Vaginitis
Keywords: Pregnancy Malaria; Bacterial Vaginoses; Trichomonas Vaginitis; Zambia; Intermittent Preventive Treatment in Pregnancy (IPTp); Sulfadoxine-Pyrimethamine; Dihydroartemisinin-Piperaquine; Metronidazole; Sub-Saharan Africa
MeSH Terms: conditions — Vaginosis, Bacterial; Trichomonas Vaginitis | interventions — Metronidazole; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Partially placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IPTp-SP plus MTZ placebo (control) (Placebo Comparator): 3 tablets each containing 500mg sulphadoxine and 25mg pyrimethamine and metronidazole placebo administered as directly observed therapy.
  Interventions: Drug: IPTp-sulphadoxine-pyrimethamine
- IPTp-SP plus MTZ (Active Comparator): 3 tablets each containing 500mg sulphadoxine and 25mg pyrimethamine and 4 tablets each containing 500mg metronidazole administered as directly observed therapy .
  Interventions: Drug: IPTp-sulphadoxine-pyrimethamine plus metronidazole
- IPTp-DP plus MTZ (Active Comparator): 3 tablets of 40mg of dihydroartemisinin and 320mg of piperaquine, first dose and will be administered as directly observed therapy with the remaining two doses on the next two consecutive days at home. 4 tablets each containing 500mg metronidazole administered as directly observed therapy.
  Interventions: Drug: IPTp-dihydroartemisinin-piperaquine plus metronidazole

INTERVENTIONS:
Drug: IPTp-sulphadoxine-pyrimethamine plus metronidazole — Metronidazole (MTZ) is indicated for the treatment of BV and TV and is also safe to administer in the second and third trimesters of pregnancy, and its use with SP or DP may result in better birth outcomes than SP alone. Malaria parasites have developed resistance against SP and the treatment is sub-optimal at clearing malaria infection compared to dihydroartemisinin-piperaquine (DP), therapy that has a suitable profile for use in IPTp. This intervention arm can be compared to the intervention arm IPTp-DP plus MTZ to assess whether DP is superior to SP in preventing adverse birth outcomes. This intervention arm will also be compared to the IPTp-SP plus MTZ placebo arm to assess whether the combination of MTZ with IPTp-SP is superior to IPTp-SP alone in reducing adverse pregnancy outcomes.
  Other Names: Fansidar; Flagyl
  Arms: IPTp-SP plus MTZ
Drug: IPTp-dihydroartemisinin-piperaquine plus metronidazole — Metronidazole (MTZ) is indicated for the treatment of BV and TV and is also safe to administer in the second and third trimesters of pregnancy, and its use with SP or DP may result in better birth outcomes than SP alone. Malaria parasites have developed resistance against SP and the treatment is sub-optimal at clearing malaria infection compared to dihydroartemisinin-piperaquine (DP), therapy that has a suitable profile for use in IPTp. This intervention arm can be compared to the intervention arm IPTp-SP plus MTZ to assess whether DP is superior to SP in in reducing adverse pregnancy outcomes.
  Other Names: Flagyl; D-ARTEPP®
  Arms: IPTp-DP plus MTZ
Drug: IPTp-sulphadoxine-pyrimethamine — The World Health Organization (WHO) recommends providing intermittent preventive treatment (IPTp) using sulphadoxine-pyrimethamine (SP) to pregnant women during the second and third trimesters of pregnancy to clear placental infection.
  Other Names: Fansidar
  Arms: IPTp-SP plus MTZ placebo (control)

SUMMARY:
Malaria in pregnancy has devastating consequences for mother and foetus. WHO recommends intermittent preventive treatment in pregnancy (IPTp) with sulphadoxine-pyrimethamine (SP) for asymptomatic women, but high-level parasite resistance to SP threatens its efficacy. Dihydroartemisinin-piperaquine (DP) has the potential to replace SP for IPTp. However, the DP strategy has not been found to be superior to SP for reducing the incidence of low birthweight (LBW), small-for-gestational age (SGA), or preterm birth. This may be the result of sulphadoxine having antibacterial properties; it is derived from sulphonamide, which have been used for decades to treat curable STIs/RTIs. However, SP is unlikely to be curative of STIs/RTIs, nor highly effective against malaria parasites. Thus, combination treatment that contains a more efficacious antimalarial and a more efficacious anti-STI/RTI may produce better birth outcomes. The investigators will therefore determine whether combining SP with metronidazole (MTZ) or, separately, DP with MTZ can improve birth outcomes more than SP alone, potentially paving the way for integrated control strategies that will reduce the dual burden of malaria and curable STIs/RTIs.

This is an individually-randomized, 3-arm, partially-placebo controlled superiority trial comparing the efficacy, safety and tolerance of IPTp-SP versus IPTp-SP with MTZ, or IPTp-DP with MTZ to reduce adverse birth outcomes attributable to malaria and curable STIs/RTIs in 5,436 women in the Nchelenge District of Zambia.

DETAILED DESCRIPTION:
Title: Effects of metronidazole plus intermittent preventive treatment of malaria in pregnancy on birth outcomes: a randomised controlled trial in Zambia.

Short Title: The ASPIRE Trial - Aiming for Safe Pregnancies by Reducing Malaria and Infections of the Reproductive Tract

Background and rationale: Current interventions in sub-Saharan Africa to reduce the burden of malaria infection and curable STIs/RTIs in pregnancy are inadequate. Malaria infection during pregnancy is responsible for 20% of all stillbirths and 11% of neonatal deaths and is strongly associated with low birthweight (LBW), preterm birth, and small-for-gestational-age (SGA) babies. To protect against adverse pregnancy outcomes in malaria-endemic areas, the WHO recommends providing IPTp-SP to pregnant women at each scheduled ANC visit as directly observed therapy from the second trimester to delivery with at least one month between doses. However, the loss of parasite sensitivity to SP has compromised the efficacy of IPTp.

Apart from syphilis and HIV screening, the WHO recommends the syndromic management of curable STIs/RTIs in low- and middle-income countries involving diagnostic and treatment algorithms based on self-reported symptoms. BV and TV are included in these guidelines. However, syndromic management fails to detect the majority of infections in women for whom STIs/RTIs are most often asymptomatic. This is of genuine consequence in pregnancy. BV is the most common urogenital disorder in the world among women of reproductive age and increases the odds of preterm delivery 1.5-2 times. TV is the most prevalent curable STI in the world and increases the odds of preterm delivery 1.5 times. BV and TV both double the odds of LBW. Although vertical transmission of TV is uncommon, maternal treatment may prevent respiratory or genital infection of the newborn. These adverse pregnancy outcomes could be averted with metronidazole (MTZ); 2g is safe and curative of TV and reduces the recurrence of BV. Importantly, the dose can be provided as directly observed therapy during ANC to ensure compliance.

IPTp-DP is the leading candidate to replace IPTp-SP. A trial in Kenya showed that IPTp-DP was superior to IPTp-SP in preventing clinical malaria episodes and other malaria-related endpoints. Alongside the trial, the investigators will conduct sub-studies that will generate important data about the mechanisms of IPTp-SP action against malaria, BV and TV.

Primary objective: To determine if IPTp with SP or DP, combined with MTZ, for the control of malaria and STIs/RTIs in pregnancy is safe and superior to IPTp with SP alone for reducing adverse pregnancy outcomes.

Hypothesis: IPTp with SP or DP, combined with MTZ, is superior to IPTp with SP alone in preventing adverse pregnancy outcomes.

Overview Study Design: A 3-arm, parallel, partially placebo-controlled, individually randomised, phase-3, superiority trial involving 5,436 (1,812 per arm) pregnant women in ANC facilities of the Nchelenge District of Zambia.

An economic evaluation will be carried out alongside the trial to estimate the cost and cost-effectiveness of interventions. In addition, the acceptability of therapy and the trade-offs between different attributes of the trial arms will be assessed using a discrete choice framework among trial participants and health care providers.

Sub-study 1: Effect of treatment on vaginal and intestinal microbiome and maternal cytokines

Objective: To characterise the effect of treatment across trial arms on the vaginal and intestinal microbiota communities, vaginal and intestinal bacterial loads and soluble markers of inflammation.

Sub-study 2: In vitro testing of sulphadoxine and other antimicrobial agents (Ndola, Zambia)

Objective: To measure the drug sensitivity of several pathogens implicated with WHO syndromes of vaginal discharge, lower abdominal pain, or genital ulcers in the presence of sulphadoxine and other antimicrobial agents.

Sites: The study will be conducted ANC facilities of the Nchelenge District of Zambia where the prior pregnancy cohort was previously carried out, malaria transmission is high, parasite resistance to SP is high, and there is a high prevalence of TV and BV among pregnant women at antenatal care facilities.

Study Population: HIV-negative pregnant women (all gravidae) between 16 and 28 weeks' gestation, as assessed by ultrasound dating who have not yet started IPTp during the current pregnancy.

Study Interventions:

Group 1: IPTp-SP plus MTZ placebo* (control) Group 2: IPTp-SP plus MTZ* Group 3: IPTp-DP plus MTZ*

SP = 3 tablets each containing 500mg sulphadoxine and 25mg pyrimethamine (Day 0) MTZ = 4 tablets each containing 500mg as directly observed therapy (Day 0) DP = 3 tablets of 40mg of dihydroartemisinin and 320mg of piperaquine (Days 0, 1, 2)

*MTZ placebo (Group 1) and active MTZ (Groups 2 and 3) will be co-administered with SP or DP during the enrolment visit (gestational week 16-19) and the last ANC visit prior to delivery (gestational week 30-34)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* HIV-negative
* Gestational age from Week 16 and 0 Days to Week 28 and 0 Days (measured by sonography)
* Carrying a single viable pregnancy
* Resident in the study area
* Express willingness to adhere to scheduled and unscheduled study visit procedures, and deliver at a trial facility

Exclusion Criteria:

* HIV-positive
* Carrying multiple pregnancies (twins, etc.),
* Known cardiac ailment
* Severe malformations or nonviable pregnancy observed by ultrasound
* History of receiving IPTp-SP during the current pregnancy
* Known allergy or contraindication to any of the study drugs
* Unable to give consent
* Concurrently participating in any other trial, including prior enrolment in this trial.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5436 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse pregnancy outcome | 8 months
  Composite endpoint of foetal morbidity, defined as any of the following: foetal loss (spontaneous abortion or stillbirth), singleton live births born with low birthweight (LBW), or preterm (PT) (LBW-PT), and subsequent neonatal death by day 28.

SECONDARY OUTCOMES:
Individual components of the primary outcome- adverse pregnancy outcomes | 8 months
  Prevalence of individual components of primary outcome
Foetal loss | 8 months
  Spontaneous abortion or stillbirth (binary)
Neonatal mortality | 8 months
  Death in the first 28 days of life (binary)
Low birthweight | 8 months from randomisation
  Birthweight <2.5 kg (binary)
Preterm birth | 8 months from randomisation
  Birth at <37 gestational weeks
Birth weight (continuous) | 8 months from randomisation
  Weight at birth (g)
Gestational age at delivery (continuous) | 8 months from randomisation
  Based on gestational age measured by ultrasound at enrolment (days)
Z-score for birthweight (continuous) | 8 months from randomisation
  Z-score for birthweight (g) from regional population reference
Small for gestational age (binary) | 8 months from randomisation
  Estimated as a stand-alone secondary outcome using the 10th percentile of regional reference charts on the corrected birthweight
Clinical malaria during pregnancy (binary) | 8 months from randomisation
  Clinical malaria at any point from enrolment including delivery and 28 day postpartum, both:
  * Documented fever (≥37.5°C), or recent history of fever in the past 24 hours, or other symptoms of acute illness that resulted in a woman seeking care with an unscheduled visit
  * Maternal malaria patent infection detectable by Rapid Diagnostic Test (RDT) for women with malaria symptoms only
Maternal malaria infection (binary) | 8 months from randomisation
  Malaria infection detected by PCR during pregnancy in the peripheral blood at any point during pregnancy (scheduled and unscheduled visits) from study registration, including delivery.
Any malaria at delivery (binary) | 8 months from randomisation
  Malaria infection at delivery detected in peripheral blood by PCR or placental blood by microscopy, PCR or histology (active infection)
Placental malaria infection (binary) | 8 months from randomisation
  Placental malaria detected by microscopy, PCR , or histology (active and past infection) including any Plasmodium species detected in the placental blood or biopsy tissue by either:
  * Placental incision smear microscopy (standard microscopy)
  * PCR placental blood (maternal)
  * Placental malaria by histology (active and past infection)
Congenital malaria infection (binary) | 8 months from randomisation
  Malaria infection detected in foetal cord blood of the new born at birth by standard microscopy
Placental malaria by histology (binary) | 8 months from randomisation
  * Active Infection:
    1. Chronic: pigment present and asexual parasites present
    2. Acute: pigment absent and asexual parasites present
  * Past Infection: Pigment in fibrin detected in the absence of asexual parasites.
  * Placental histology categories
    1. Any
    2. Active
    3. Active acute
    4. Active chronic
    5. Past
Placental Inflammation or chorioamnionitis (binary) | 8 months from randomisation
  Any inflammation in the placenta or chorioamnionitis detected by placental histology
Maternal anaemia (binary) and haemoglobin concentration (continuous (g/dL) at enrolment and delivery | 8 months from randomisation
  Definition:
  * No anaemia (Hb >11 g/dL)
  * Mild (Hb >10 to <11 g/dL)
  * Moderate (Hb >7 to <10 g/dL
  * Severe (Hb <7 g/dL)
Congenital anaemia in umbilical cord blood at delivery | 8 months from randomisation
  Hb<12.5 g/dL in umbilical cord blood at birth, which is 2 standard deviations below the mean cord Hb in developed countries
Congenital malformations (binary) | 8 months from randomisation
  Physical abnormality of live born baby detected at delivery or newly noted abnormality during the infant visits (7 days or 2-6 weeks post-natal)
Maternal mortality (binary) | 8 months from randomisation
  Maternal mortality from registration until 28 days after delivery
SAEs and AEs defined by MedDRA (listings) | 8 months from randomisation
  AEs and SAEs will be defined according to the Medical Dictionary for Regulatory Activities (MedDRA) and reported by study arm:
  * Overall
  * By system organ class and preferred term
History of vomiting study drug - Prevalence at each cycle of treatment (binary) | 8 months from randomisation
  Vomited within 30 minutes of taking study drug at any scheduled administration
Dizziness - Prevalence at each cycle of treatment | 8 months from randomisation
  Dizziness at any point within 30 minutes of first drug administered during a treatment cycle, reported as Mothers adverse event
Gastrointestinal complaints - Prevalence at each cycle of treatment (binary) | 8 months from randomisation
  Nausea or vomiting within 30 minutes of first drug administered during a treatment cycle
Presence of any one or more STIs/RTIs - Prevalence at enrolment (binary) | 8 months from randomisation
  Any or more infection of syphilis, gonorrhoea, chlamydia, trichomoniasis, and bacterial vaginosis

CONTACTS AND LOCATIONS:
Overall Officials: R. Matthew Chico, MPH, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Nchelenge District Health Facilites, Nchelenge, Luapula Province, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon receiving formal request and subject to sharing agreement.
Supporting Information: Study Protocol
Time Frame: Five years
Access Criteria: The full protocol will be available on request to any interested professional. All requests for data for secondary analysis will be considered by a Data Access Committee to ensure that use of data is within the terms of consent and ethics approval.